CLINICAL TRIAL: NCT04959747
Title: Acupuncture for Olfactory Dysfunction in Infected COVID-19 Patients: A Randomized, Sham-controlled Clinical Trial
Brief Title: Acupuncture for Olfactory Dysfunction in Infected COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Tseung Kwan O Hospital, Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Acupuncture for OD
Record Dates: First submitted 2021-07-12; First posted 2021-07-13 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Olfactory Dysfunction; Covid19
Keywords: olfactory dysfunction; acupuncture; COVID-19; randomized; sham controlled trial
MeSH Terms: conditions — COVID-19 | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: single blinded, randomized sham controlled, cross-over clinical trial
Who Masked: Participant
Masking Description: Subjects of both groups will be randomly assigned into 2 groups, the acupuncture group or the control (sham) acupuncture group with 1:1 ratio. For randomization, simple, complete non-sequential random numbers will be generated in advance by a computer program in a block of four, and kept by the principal investigator. After a patient's eligibility is confirmed, a randomization number which corresponds to the group allocation will be provided to the acupuncturist by the PI. This arrangement will ensure that the clinical assessor and participants are blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental): Subject will be scheduled for a total of 8 sessions of acupuncture treatment, to be done by the 30 minutes for each session, twice per week over a 4-week period.
  Body acupuncture will choose eight acupoints as Yingxiang (LI20),Shangxing (GV23), BiTong, Yintang, Hegu. Disposable acupuncture needle (0.25 mm in diameter and 25-30mm in length) are inserted at a depth of 10-25 mm obliquely into scalp acupuncture points (ShangXing, YinTang) and straightly into face/body acupuncture points (Yingxiang, BiTong, Hegu).
  We will also deliver electro-acupuncture will be applied to the face points at fast and dispersed waves through electric needle stimulator which is provided by Chinese Medicine Clinic (ES-160 6-Channel Programmable electro-acupuncture) for 30 minutes.
  Interventions: Other: acupuncture
- sham-acupuncture group (Placebo Comparator): For subjects assigned to control group, Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2" / 0.30 x 30 mm) will be applied to serve as sham control at the same acupoints with the same stimulation modality, except that the needles are only adhered to the skin instead of insertion. Its validity and credibility have been well demonstrated.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Body acupuncture will choose eight acupoints as Yingxiang (LI20),Shangxing (GV23), BiTong, Yintang, Hegu. Disposable acupuncture needle (0.25 mm in diameter and 25-30mm in length) are inserted at a depth of 10-25 mm obliquely into scalp acupuncture points (ShangXing, YinTang) and straightly into face/body acupuncture points (Yingxiang, BiTong, Hegu).
  We will also deliver electro-acupuncture will be applied to the face points at fast and dispersed waves through electric needle stimulator which is provided by Chinese Medicine Clinic (ES-160 6-Channel Programmable electro-acupuncture) for 30 minutes.

SUMMARY:
In this a 12-week, single blinded, randomized sham controlled, and cross-over clinical trial. It will be conducted to explore the safety and efficacy of acupuncture for olfactory dysfunction in infected COVID-19 patients in Hong Kong.

DETAILED DESCRIPTION:
This is a single blinded, randomized sham controlled, and cross-over clinical trial. 40 Post COVID-19 patients presenting to olfactory dysfunction will be recruited. 40 patients will be randomly assigned into 2 groups, the acupuncture group (AC) and the sham acupuncture group (SAC) with 1:1 ratio, for 4-week treatment and 2-week follow-up. After the follow-up, the sham group will be conducted with real acupuncture for another 4 weeks and the real acupuncture group will be conducted with the 4-week sham acupuncture.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been previously diagnosed to be infected with COVID-19 and are discharged from local hospitals with all the follows: 1) post COVID-19 olfactory dysfunction with moderate or severe grades (base on UPSIT-TC scores, the cutoff scores are set at 29.5 for male and 30.5 for female); 2) post COVID-19 olfactory dysfunction who did not undergo treatment; 3) no history of trauma, injury or surgery to head or nose or any bleeding from the nose; 4) aged 18 to 80 years who are able to read and write Chinese.

Exclusion Criteria:

Patients will be excluded if they have one or more of follows: 1) patients with olfactory or gustatory dysfunctions before the COVID-19 epidemic; 2) patients with history of chronic rhinosinusitis or nasal polyposis; 3) history of nasal surgery (including rhino/septoplasty with or without functional endoscopic sinus surgery; 4) Pregnant or breastfeeding women.; 5) Medical history: cancers, conditions that affect the nervous system, such as Parkinson's disease or Alzheimer's disease, and/or any other serious diseases; 6) Unstable medical conditions; 7) Patients who have received acupuncture treatment within one month, 8) Alcoholism or drug abuse in past 1 year; 9) Have needle phobia; 10) Have known history of developing acupuncture related severe adverse reaction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
ASOF scores | 1, 6, 8, 12, 14 weeks
  The Assessment of Self-reported Olfactory Functioning and olfaction related quality of life (ASOF) is a 12-item validated questionnaire, it can be subdivided into three domains: the one-item subjective olfactory capability scale (SOC), the five-item self-reported capability of perceiving specific odors scale (SRP), and the six-item olfactory-related quality of life (ORQ) scale. We proceeded to calculate cutoff scores for the three scales. Patients will be considered to have abnormal olfactory capabilities if the SOC score was equal to or less than 3. Scale from 10 (best possible) to 0 (worst possible-unable to smell). Patients were considered to have problems smelling odors if the SRP score was equal to or less than 2.9 (Scale from 0 to 5) Patients were considered to have smell-related problems in quality of life if the ORQ score was equal to or less than 3.7 (Scale from 0 to 6)
sQOD-NS scores | 1, 6, 8, 12, 14 weeks
  The Short version of the Questionnaire of Olfactory Disorders-Negative Statements (sQOD-NS) is a 7-item patient-reported outcome questionnaire. Patients rated the item proposition from 0 (agree) to 3 (disagree) with total score ranging from 0 (significant impact of olfactory dysfunction on quality of life) to 21 (no impact on quality of life). The sQOD-NS is composed of seven questions including social, eating, annoyance, and anxiety and assessed using a 4-point Likert scale (0-3). A higher score means better olfactory specific quality of life.

SECONDARY OUTCOMES:
UPSIT-TC | 0, 14 weeks
  The University of Pennsylvania Smell Identification Test (UPSIT) is widely used internationally and the worldwide standard for olfactory testing. UPSIT is a 40-item "scratch and sniff" multiple choice test to assess how well participants can identify different odors. Patients will be required to identify each of the 40 odors from four alternatives listed for each odor. The number of correct responses provided a test score such that patients could be categorized into one of four categories: mild, moderate, severe, or total loss. The test is scored by the number of odors identified correctly to generate a maximum score of 40.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fung CHO, Dr., Principal Investigator — Department of Medicine, Tseung Kwan O Hospital
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The sharing of the research data of individual participants will be available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be shared within 7 years of the completion of this study.
Access Criteria: By requirement